CLINICAL TRIAL: NCT05020899
Title: Quit For Life (QFL): Smoking Cessation Among Chinese Smokers Living With HIV
Acronym: QFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-41807; 1R21CA243835-01A1 (NIH)
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Smoking Cessation; HIV Infections
Keywords: Quit for Life (QFL); Smoking cessation counselors; WeChat messages; Nicotine replacement therapy; Self-help smoking cessation guide; People living with HIV/AIDS (PLH)
MeSH Terms: conditions — Smoking Cessation; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quit for Life group (Experimental): Participants randomized to this arm will receive a 8 week quit smoking program delivered by trained counselors and messages to their cell phones. Participants will also be offered nicotine replacement therapy (gum or patch, depending on which one is available) and a self-help guide with information about quitting smoking.
  Interventions: Behavioral: Sessions with a trained counselor; Other: Cell phone messages; Other: Offered nicotine replacement therapy; Other: Self-help guide for quitting smoking
- Control group (Active Comparator): Participants randomized to this arm will be offered nicotine replacement therapy (gum or patch, depending on which one is available) and a self-help guide with information about quitting smoking.
  Interventions: Other: Offered nicotine replacement therapy; Other: Self-help guide for quitting smoking

INTERVENTIONS:
Behavioral: Sessions with a trained counselor — 4 sessions will be provided with a trained counselor who will discuss the participant's' smoking habits with them and strategies to help them quit. The first session is in-person, lasts for 20 minutes, and typically happens when the participant comes to the HIV clinic to pick up their medication. Sessions 2 through 4 are over the telephone and last for 15 minutes each. These occur 1 week, 4 weeks, and 8 weeks after the first session.
  Arms: Quit for Life group
Other: Cell phone messages — Brief messages that give tips to help quit smoking will be sent to participants' cell phones using WeChat. 3 messages per day will be sent for the first week, 2 messages per day for the next 3 weeks, 1 message per day for the next 1 week, and 1-2 messages per week for the rest of the time
  Arms: Quit for Life group
Other: Offered nicotine replacement therapy — Participants will be offered nicotine replacement therapy (gum or patch, depending on which one is available).
Other: Self-help guide for quitting smoking — Participants will be offered a self-help guide with information about quitting smoking.

SUMMARY:
The purpose of this two arm randomized clinical trial (RCT) is to test if a smoking cessation program called Quit for Life (QFL) which was developed by the investigators is effective for patients in China with HIV who smoke. This program is designed to suit the needs of people with HIV who smoke in China.

Eligible participants who provide consent will be randomized into either the QFL or the Control group.

The QFL group will receive a quit smoking program that lasts for 8 weeks with two parts-

1. 4 sessions with a trained counselor who will discuss the participants' smoking habits and strategies to help them quit.
2. Messages sent to the participants' cell phone using WeChat.

The Control group will not have sessions with a trained counselor or receive messages sent to their cell phone.

Both groups will be offered nicotine replacement therapy and a self-help guide with information about quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive (by being at the HIV clinic and receiving care)
* Receiving ART treatment from the clinic (by being at the HIV clinic and receiving care)
* Smokes ≥ 5 cigarettes per day
* Able to speak and read in Mandarin Chinese
* Self-reported anticipate to receive ART treatment from the clinic for at least 9 months
* Own a cell phone
* Be willing to set a quit date within 1 month after baseline assessment

Exclusion Criteria:

* Self-reported using other smoking cessation program or medication
* Having a serious health problem that may make them unsuitable to stay in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Quintiliani, PhD, Principal Investigator — Boston Medical Center; Hao Liang, PhD, Principal Investigator — Guangxi Medical University
Locations (2):
- Boston Medical Center, Boston, Massachusetts, United States
- Guangxi Medical University, Guangxi, Nanning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Yang S, Xie Z, Guo B, Lan Y, Li Y, Jiang Y, Forman LS, Lunze K, Liang B, Abdullah AS, Ye L, Liang H, Quintiliani LM. WeChat-based Messaging and Behavioral Counseling for Smoking Cessation for People with HIV in China: a Randomized Controlled Pilot Trial. AIDS Behav. 2025 Dec;29(12):3866-3876. doi: 10.1007/s10461-025-04823-7. Epub 2025 Jul 24. PMID 40705206

RESULTS

PARTICIPANT FLOW:
Period: 8 Week Follow-up
Arm/Group | Quit for Life Group | Control Group
Started | 54 | 55
Completed | 51 | 49
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6
Period: 12 Week Follow-up
Arm/Group | Quit for Life Group | Control Group
Started | 51 | 49
Completed | 50 | 48
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quit for Life Group | Control Group | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (15) | 46 (16) | 45 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 52 | 53 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 54 | 55 | 109
Region of Enrollment [Number; unit: participants]
  China | 54 | 55 | 109
Cigarettes Smoked in the Previous 30 Days [Mean (Standard Deviation); unit: cigarettes] | 502.2 (242.3) | 579.3 (218.0) | 541.1 (232.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically Verified Smoking Cessation
Description: Defined as not smoking during the previous 7 days, not even a puff, validated by measuring CO level (<8ppm) in the exhaled air
Time Frame: 12 weeks
Population: Data are missing for 6 participants in the Quit for Life group and 9 participants in the Control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 44 | 39
Participants | 26 | 10

2. Secondary Outcome: Number of Participants That Self Reported Smoking Cessation at 8 Weeks
Description: Participants will report if they did not smoke in the previous 7 days by answering questions in an interviewer-administered questionnaire.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 51 | 49
Participants | 29 | 37

3. Secondary Outcome: Number of Participants That Self Reported Smoking Cessation at 12 Weeks
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 50 | 48
Participants | 29 | 40

4. Secondary Outcome: Change in Number of Cigarettes Smoked in the Previous 30 Days at 8 Weeks
Description: Participants will report the number of cigarettes they smoked in the previous 30 days by answering questions in an interviewer-administered questionnaire.
Time Frame: baseline, 8 weeks
Population: Data are missing for 23 participants in the Quit for Life group and 13 participants in the Control group.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 28 | 36
cigarettes | -169.29 (287.08) | -170.83 (163.66)

5. Secondary Outcome: Change in Number of Cigarettes Smoked in the Previous 30 Days at 12 Weeks
Description: as for outcome 4
Time Frame: baseline, 12 weeks
Population: Data are missing for 24 participants in the Quit for Life group and 10 participants in the Control group.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 26 | 38
cigarettes | -208.85 (263.93) | -191.84 (175.42)

6. Secondary Outcome: Number of Quit Attempts at 8 Weeks
Description: Participants will report the number of quit attempts since the study started by answering questions in an interviewer-administered questionnaire.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 51 | 49
Participants
  No attempts | 7 | 13
  1 or more attempts | 44 | 36

7. Secondary Outcome: Number of Quit Attempts at 12 Weeks
Description: as for outcome 6
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 50 | 48
Participants
  No attempts | 1 | 10
  1 or more attempts | 49 | 38

8. Secondary Outcome: Adherence to Antiretroviral Treatments (ART) at 8 Weeks
Description: ART adherence will be assessed with the investigator developed, interviewer-administered 'Adherence to HIV medicine' questionnaire. This questionnaire assesses degree of adherence to taking HIV medicine on time by selecting a number between 0 and 10, where 0 = never on time [worse outcome] and 10 = always on time [best outcome]. Higher scores are more favorable.
Time Frame: 8 weeks
Population: Data are missing for 1 participant in the Control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 51 | 48
units on a scale | 9.65 (0.59) | 9.10 (1.79)

9. Secondary Outcome: Adherence to Antiretroviral Treatments (ART) at 12 Weeks
Description: as for outcome 8
Time Frame: 12 weeks
Population: Data are missing for 1 participant in the Control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 50 | 47
units on a scale | 9.42 (1.43) | 9.02 (2.20)

10. Secondary Outcome: Quality of Life (QOL) in the Dimensions of Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression at 12 Weeks
Description: The EuroQol- 5 Dimension (EQ-5D) will be used to assess QOL. It is a questionnaire with five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a scale of 0 to 100 where 0 means the worst health and 100 means the best health the participant can imagine.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 50 | 48
units on a scale | 83.90 (9.81) | 79.75 (9.90)

11. Other Pre Specified Outcome: Intervention Satisfaction at 8 Weeks
Description: Participant satisfaction with the intervention will be assessed using an investigator-developed questionnaire
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 51 | 49
Participants
  Met all of your goal | 17 | 11
  Met some/none of your goal | 34 | 38

12. Other Pre Specified Outcome: Intervention Satisfaction at 12 Weeks
Description: Participant satisfaction with the intervention will be assessed using an investigator-developed questionnaire
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Quit for Life Group | Control Group
Number analyzed (Participants) | 50 | 48
Participants
  Met all of your goal | 21 | 8
  Met some/none of your goal | 29 | 40

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Quit for Life Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/54 | 1/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 0/54 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05020899/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT05020899/ICF_001.pdf